CLINICAL TRIAL: NCT03845491
Title: ASSIST Registry to Assess the Procedural Success and Clinical Outcomes Associated With Various Operator Techniques for Mechanical Thrombectomy in Large Vessel Occlusions (LVO).
Brief Title: ASSIST Registry Studying Various Operator Techniques
Status: Completed | Type: Observational
Sponsor: Stryker Neurovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: CDM10001414
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- SR Classic: SR (Trevo®]) + BGC (FlowGate2] or Merci)
  Interventions: Device: Mechanical Thrombectomy
- SR Combination: SR (Trevo) + Asp Cath (AXS Catalyst DAC, Vecta) ± Pump + LS (AXS Infinity LS, AXS Infinity LS Plus)
  or
  SR (Trevo) + Asp Cath (AXS Catalyst DAC) ± Pump + BGC (FlowGate2 or Merci)
  Interventions: Device: Mechanical Thrombectomy
- Direct Aspiration: Asp Cath (AXS Catalyst DAC, Vecta) ± Pump + LS (AXS Infinity LS, AXS Infinity LS Plus)
  or
  Asp Cath (AXS Catalyst DAC) ± Pump + BGC (FlowGate2, Merci)
  Interventions: Device: Mechanical Thrombectomy

INTERVENTIONS:
Device: Mechanical Thrombectomy — Treatment of LVO with mechanical thrombectomy

SUMMARY:
The purpose of this Registry is to assess the procedural success and clinical outcomes associated with various operator techniques for mechanical thrombectomy in large vessel occlusions (LVO).

DETAILED DESCRIPTION:
ASSIST is a prospective, global, consecutive enrollment Registry of anterior circulation acute ischemic stroke patients with an LVO who undergo treatment with one of the interventional techniques using Stryker Neurovascular devices for the first pass. The purpose of this Registry is to assess the procedural success and clinical outcomes associated with various operator techniques for mechanical thrombectomy in large vessel occlusions (LVO) in the anterior circulation. Data will be collected on the use of Stryker market-released neurovascular mechanical access and mechanical thrombectomy devices that are commercially available or that may be approved for commercial use during the conduct of the Registry. This Registry will also collect data, including time-to-treatment and quality of life measures, to allow for subset analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who experienced acute ischemic stroke (AIS), eligible for restoration of blood flow using Stryker Neurovascular market-released products in the neurovasculature to remove thrombus
2. Occlusion of intracranial anterior circulation vessel
3. Subject or subject's legally authorized representative (LAR) has signed the informed consent form prior to or within 48 hours post-procedure
4. Subject is willing to comply with the protocol follow-up requirements
5. The intended technique and treated technique must be one of the following techniques for the first thrombectomy pass in the neurovasculature per Instructions For Use (IFU): Technique Category/Devices: SR Classic/SR + BGC, SR Combination/SR + Asp Cath ± Pump + BGC or LS, Direct Aspiration/Asp Cath ± Pump + BGC or LS,

Exclusion Criteria:

The subject is participating in another device trial or any other clinical trial where the study procedure or treatment might confound this study's endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects experiencing acute ischemic stroke (AIS) who are eligible for restoration of blood flow using Stryker Neurovascular market-released products in the neurovasculature to remove thrombus
Sampling Method: Probability Sample
Enrollment: 1492 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2023-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rishi Gupta, MD, Principal Investigator — WellStar Medical Group; Markus Möhlenbruch, MD, Principal Investigator — University Hospital Heidelberg
Locations (72):
- United States (38):
  - Banner Desert, Mesa, Arizona
  - Kaiser Permanente Fontana, Fontana, California
  - Kaiser Permanente LA, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Doctors Medical Center Modesto, Modesto, California
  - UC Irvine, Orange, California
  - Dignity Health/ Mercy San Juan, Rancho Cordova, California
  - Stanford, Stanford, California
  - St. Mary's Medical Center, Delray Beach, Florida
  - Memorial Healthcare System, Hollywood, Florida
  - Baptist Jacksonville, Jacksonville, Florida
  - University of S. Florida/Tampa General, Tampa, Florida
  - WellStar Health System/ Kennestone Hospital, Marietta, Georgia
  - Advocate Hospital, Oak Lawn, Illinois
  - Indiana University, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - UMASS, Worcester, Massachusetts
  - McLaren Regional Medical Facility, Flint, Michigan
  - Sparrow Health, Lansing, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Buffalo University, Buffalo, New York
  - Mount Sinai, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - Riverside Methodist- OHRI, Columbus, Ohio
  - Mercy St. Vincent, Toledo, Ohio
  - University of Oklahoma Medical Center (OU - OKC), Oklahoma City, Oklahoma
  - Legacy Emanuel Medical Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - MUSC, Charleston, South Carolina
  - Semmes Murphey Foundation, Memphis, Tennessee
  - University Medical Center- El Paso, El Paso, Texas
  - Valley Baptist Harlingen, Harlingen, Texas
  - West Virginia University Hospital, Morgantown, Virginia
  - Aurora St. Luke's, Milwaukee, Wisconsin
- Belgium (2):
  - Ghent University Hospital, Ghent
  - AZ Sint-Jan AV Brugge Oostende, Ostend
- Toronto Western Hospital, Toronto, Canada
- Hradec Kralove, Hradec Králové, Czechia
- France (4):
  - CHU Bordeaux_GH Pellegrin, Bordeaux
  - Hospital Cavale Blanche CHU Brest, Brest
  - CHU Lyon- Hopital P. Wertheimer, Bron
  - CHU Rouen, Rouen
- Germany (6):
  - Klinikum Dortmund, Dortmund
  - University Hospital Heidelberg, Heidelberg
  - Klinikum Kassel, Kassel
  - Klinikum Rechts Der Isar, Munich
  - Klinikum LMU, Munich
  - Klinikum Vest Recklinghausen, Recklinghausen
- Italy (6):
  - Ospedale Policlinico san Martino, Genova
  - AOPU G. Martino, Messina
  - AO Parma, Parma
  - AO San Camillo Forlanini, Roma
  - Azienda Ospedaliera Siena, Siena
  - AO Modena, Via Giardini
- South Korea (2):
  - Cheonnam University Hospital, Gwangju
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon
- Spain (8):
  - Hospital Clínico Universitario de Valladolid, Valladolid, Castille and León
  - Hospital Universitario Central de Asturias - HUCA, Oviedo, Vigo
  - Hospital Vall de Hebron, Barcelona
  - Hospital de la Princesa, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Son Espases de Mallorca, Palma de Mallorca
  - Hospital Universitario Marqués de Valdecilla, Santander
- Switzerland (3):
  - University Hospital Basel, Basel
  - HUG Geneva, Geneva
  - CHUV, Lausanne
- Charing Cross, London, United Kingdom

REFERENCES:
- [Derived] Molaie A, Miralbes S, Naravetla B, Spiotta AM, Loehr C, Martinez-Galdamez M, McTaggart RA, Defreyne L, Vega P, Zaidat OO, Jenkins P, Mohlenbruch M, Gupta R, Liebeskind DS; ASSIST Investigators. Incomplete reperfusion and the presence of distal emboli in predicting clinical outcome after endovascular thrombectomy. BMJ Surg Interv Health Technol. 2025 Apr 10;7(1):e000345. doi: 10.1136/bmjsit-2024-000345. eCollection 2025. PMID 40226203
- [Derived] Luff MK, Khezri N, Miralbes S, Naravetla B, Spiotta AM, Loehr C, Martinez-Galdamez M, McTaggart RA, Defreyne L, Vega P, Zaidat OO, Price LL, Gupta R, Mohlenbruch MA, Liebeskind DS; ASSIST Investigators. Hemorrhagic transformation in acute ischemic stroke: hemorrhagic subtypes and symptomatic intracranial hemorrhage. J Neurointerv Surg. 2025 Jun 16;17(7):673-682. doi: 10.1136/jnis-2024-021725. PMID 38969497

RESULTS

PARTICIPANT FLOW:
Groups:
- SR Combination: SR (Trevo) + Asp Cath (AXS Catalyst DAC, Vecta) ± Pump + LS (AXS Infinity LS, AXS Infinity LS Plus)
  or
  SR (Trevo) + Asp Cath (AXS Catalyst DAC) ± Pump + BGC (FlowGate2 or Merci)
  Mechanical Thrombectomy: Treatment of LVO with mechanical thrombectomy
- Direct Aspiration: Asp Cath (AXS Catalyst DAC, Vecta) ± Pump + LS (AXS Infinity LS, AXS Infinity LS Plus)
  or
  Asp Cath (AXS Catalyst DAC) ± Pump + BGC (FlowGate2, Merci)
  Mechanical Thrombectomy: Treatment of LVO with mechanical thrombectomy
Period: Overall Study
Arm/Group | SR Classic | SR Combination | Direct Aspiration
Started | 247 | 697 | 548
Completed | 209 | 563 | 432
Not Completed | 38 | 134 | 116

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SR Classic | SR Combination | Direct Aspiration | Total
Number analyzed (Participants) | 247 | 697 | 548 | 1492
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 1 | 1
  Between 18 and 65 years | 66 | 191 | 192 | 449
  >=65 years | 181 | 506 | 355 | 1042
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.4 (14.3) | 71.8 (13.1) | 68.1 (15.4) | 70.4 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 379 | 281 | 781
  Male | 126 | 318 | 267 | 711
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 12 | 2 | 15
  South Korea | 20 | 33 | 11 | 64
  Belgium | 14 | 45 | 3 | 62
  United States | 47 | 327 | 280 | 654
  Czechia | 20 | 16 | 4 | 40
  Italy | 1 | 42 | 52 | 95
  United Kingdom | 0 | 0 | 1 | 1
  France | 0 | 17 | 2 | 19
  Switzerland | 0 | 45 | 8 | 53
  Germany | 0 | 115 | 52 | 167
  Spain | 144 | 45 | 133 | 322

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieved Good Functional Outcome (mRS 0-2) at Day 90
Description: This measure assesses clinical outcome using the Modified Rankin Scale (mRS). Modified Rankin Scale measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It is a score ranging from 0-6 with the following degree of disability: 0 = No symptoms at all; no limitations and no symptoms; 1 = No significant disability, 2 = Slight disability; 3 = Moderate disability; 4 = Moderate severe disability, 5 = Severe disability; 6= Death. The lower mRS Score indicates less disability, and higher score indicates increased disability.
Time Frame: 90 Days (±14 days)
Population: Available mRS scores at 90Days (±14 days) of the enrolled population
Measure: Count of Participants; unit: Participants
Arm/Group | SR Classic | SR Combination | Direct Aspiration
Number analyzed (Participants) | 237 | 666 | 506
Participants | 140 | 351 | 273

2. Primary Outcome: Percentage of Subjects Achieved eTICI 2c or Greater on First Pass (Adjudicated by the Core Lab)
Description: This outcome measures percentage of subjects who achieved complete reperfusion after the first pass, defined by eTICI score of 2c or greater. Independent Imaging Core Lab adjudicated the outcome using the Expanded Treatment in Cerebral Infarction (eTICI) scale. The higher eTICI score indicates successful revascularization.
  The Expanded TICI (eTICI) Perfusion Score Categories are:
  * 0: Equivalent to no reperfusion or 0% filling of the downstream territory
  * 1: Reflects thrombus reduction without any reperfusion of distal arteries
  * 2a: Reperfusion in less than half or 1-49% of the territory
  * 2b50: 50-66% reperfusion
  * 2b67: 67-89% reperfusion
  * 2c: 90-99% reperfusion
  * 3: Complete or 100% reperfusion
Time Frame: At the time of procedure, after the first pass
Population: Available core lab adjudicated procedural endpoint data of the enrolled subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | SR Classic | SR Combination | Direct Aspiration
Number analyzed (Participants) | 233 | 680 | 529
Participants | 110 | 309 | 193

3. Secondary Outcome: Percentage of Subjects With an Excellent Functional Outcome at Day 90
Description: Percentage of subjects with an excellent functional outcome of mRS of 0-1 at Day 90 (± 14).
  Modified Rankin Scale measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It is a score ranging from 0-6 with the following degree of disability: 0 = No symptoms at all, no limitations and no symptoms; 1 = No significant disability, 2 = Slight disability; 3 = Moderate disability; 4 = Moderate severe disability, 5 = Severe disability; 6= Death. The lower mRS Score indicates less disability.
Time Frame: 90 Days (±14 days)
Measure: Count of Participants; unit: Participants
Arm/Group | SR Classic | SR Combination | Direct Aspiration
Number analyzed (Participants) | 237 | 666 | 506
Participants | 112 | 264 | 209

4. Secondary Outcome: Percentage of Subjects With an "Early Response" Defined by NIHSS Score
Description: Percentage of subjects with an "early response" at Discharge/Day5-7 (whichever is earlier) defined as a NIHSS drop of ≥10 points from baseline or NIHSS score of 0 or 1.
  NIHSS (National Institutes of Health Stroke Scale) is an assessment to objectively quantify the impairment caused by a stroke. It is composed of 11 items, each of which scores a specific ability. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
Time Frame: Discharge/ Day 5-7 (Whichever is earlier)
Measure: Count of Participants; unit: Participants
Arm/Group | SR Classic | SR Combination | Direct Aspiration
Number analyzed (Participants) | 236 | 646 | 507
Participants | 156 | 376 | 294

5. Secondary Outcome: Quality of Life at Day 90 Based on EQ5D5L Score
Description: The Euro Quality of Life Questionnaire - 5 Level 5D Version (EQ5D5L) is composed of 5 dimensions- mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is evaluated by the subject on 5 level scale: no problems, slight problems, moderate problems, severe problems and extreme problems. The outcome reported shows severe and extreme levels were combined and only 4 levels are reported.
Time Frame: Day 90 (±14 days)
Population: The analysis population is based on availability of the self reported data
Measure: Count of Participants; unit: Participants
Arm/Group | SR Classic | SR Combination | Direct Aspiration
Number analyzed (Participants) | 182 | 492 | 384
Participants
  Mobility:: No Problems | 103 | 247 | 187
  Mobility:: Slight Problems | 36 | 94 | 77
  Mobility:: Moderate Problems | 22 | 68 | 56
  Mobility:: Severe/Extreme Problems | 21 | 83 | 64
  Self-care:: No Problems | 116 | 293 | 227
  Self-care:: Slight Problems | 30 | 70 | 68
  Self-care:: Moderate Problems | 19 | 53 | 38
  Self-care:: Severe/Extreme Problems | 17 | 76 | 51
  Usual Activities: No Problems | 95 | 212 | 154
  Usual Activities: Slight Problems | 44 | 107 | 96
  Usual Activities: Moderate Problems | 26 | 77 | 61
  Usual Activities: Severe/Extreme Problems | 17 | 96 | 73
  Pain/Discomfort:: number analyzed (Participants) | 182 | 491 | 384
  Pain/Discomfort:: No Problems | 110 | 261 | 205
  Pain/Discomfort:: Slight Problems | 50 | 124 | 99
  Pain/Discomfort:: Moderate Problems | 20 | 78 | 59
  Pain/Discomfort:: Severe/Extreme Problems | 2 | 28 | 21
  Anxiety/Depression:: number analyzed (Participants) | 182 | 489 | 383
  Anxiety/Depression:: No Problems | 118 | 253 | 201
  Anxiety/Depression:: Slight Problems | 41 | 125 | 107
  Anxiety/Depression:: Moderate Problems | 11 | 85 | 46
  Anxiety/Depression:: Severe/Extreme Problems | 12 | 26 | 29

6. Secondary Outcome: Percentage of Subjects Achieved eTICI 2b50, eTICI 2b67, eTICI 2c, or eTICI 3 on First Pass After Primary Technique Used and at the End of Endovascular Procedure.
Description: This outcome reports percentage of subjects who achieved eTICI 2b50, eTICI 2b67, eTICI 2c,or eTICI 3 on first pass after primary technique used and at the end of the endovascular procedure.
  Independent Imaging Core Lab adjudicated the outcome using the Expanded Treatment in Cerebral Infarction (eTICI) scale. The higher eTICI score indicates successful revascularization.
  The Expanded TICI (eTICI) Perfusion Score Categories are:
  * 0: Equivalent to no reperfusion or 0% filling of the downstream territory
  * 1: Reflects thrombus reduction without any reperfusion of distal arteries
  * 2a: Reperfusion in less than half or 1-49% of the territory
  * 2b50: 50-66% reperfusion
  * 2b67: 67-89% reperfusion
  * 2c: 90-99% reperfusion
  * 3: Complete or 100% reperfusion
Time Frame: At the time of procedure, after the first pass, and at the end of the procedure
Population: Subjects with available 90 Day core lab imaging data
Measure: Count of Participants; unit: Participants
Arm/Group | SR Classic | SR Combination | Direct Aspiration
Number analyzed (Participants) | 245 | 692 | 544
Participants
  After First Pass: number analyzed (Participants) | 233 | 680 | 529
  After First Pass: eTICI 0, 1, or 2a | 66 | 179 | 200
  After First Pass: eTICI 2b50 | 16 | 55 | 52
  After First Pass: eTICI 2b67 | 41 | 137 | 84
  After First Pass: eTICI 2c | 31 | 149 | 105
  After First Pass: eTICI 3 | 79 | 160 | 88
  At the End of Procedure: eTICI 0, 1, or 2a | 7 | 33 | 17
  At the End of Procedure: eTICI 2b50 | 2 | 38 | 36
  At the End of Procedure: eTICI 2b67 | 65 | 172 | 134
  At the End of Procedure: eTICI 2c | 57 | 238 | 200
  At the End of Procedure: eTICI 3 | 114 | 211 | 157

7. Secondary Outcome: Time From Groin Puncture to Achieve eTICI 2b50, eTICI 2b67, eTICI 2c, or eTICI 3 After the First Pass
Description: This outcome measures overall time (in minutes) observed from groin puncture to the specific eTICI reperfusion score at end of first pass for treatment of target occlusion. Each subject can only be in one eTICI category and therefore they are mutually exclusive.
  Independent Imaging Core Lab adjudicated the outcome using the Expanded Treatment in Cerebral Infarction (eTICI) scale. The higher eTICI score indicates successful revascularization.
  The Expanded TICI (eTICI) Perfusion Score Categories are:
  * 0: Equivalent to no reperfusion or 0% filling of the downstream territory
  * 1: Reflects thrombus reduction without any reperfusion of distal arteries
  * 2a: Reperfusion in less than half or 1-49% of the territory
  * 2b50: 50-66% reperfusion
  * 2b67: 67-89% reperfusion
  * 2c: 90-99% reperfusion
  * 3: Complete or 100% reperfusion
Time Frame: During the procedure, from groin puncture to after the first pass
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | SR Classic | SR Combination | Direct Aspiration
Number analyzed (Participants) | 167 | 498 | 326
Minutes
  eTICI 2b50 | 21.94 (8.5) | 23.31 (12.4) | 20.14 (13.9)
  eTICI 2b67 | 25.68 (17.0) | 28.85 (16.5) | 19.24 (12.3)
  eTICI 2c | 22.77 (11.2) | 27.59 (13.7) | 18.61 (14.0)
  eTICI 3 | 23.19 (13.6) | 27.17 (16.0) | 20.40 (10.7)

8. Secondary Outcome: Overall Time From Groin Puncture to Achieve Final Reperfusion of eTICI 2c or 3
Description: This outcome measures the overall time (in minutes) observed from groin puncture to final reperfusion of eTICI 2c or 3 for treatment of target occlusion.
  Independent Imaging Core Lab adjudicated the outcome using the Expanded Treatment in Cerebral Infarction (eTICI) scale. The higher eTICI score indicates successful revascularization.
  The Expanded TICI (eTICI) Perfusion Score Categories are:
  * 0: Equivalent to no reperfusion or 0% filling of the downstream territory
  * 1: Reflects thrombus reduction without any reperfusion of distal arteries
  * 2a: Reperfusion in less than half or 1-49% of the territory
  * 2b50: 50-66% reperfusion
  * 2b67: 67-89% reperfusion
  * 2c: 90-99% reperfusion
  * 3: Complete or 100% reperfusion
Time Frame: Time of procedure, from groing puncture to revascularization
Population: Limited to subjects who achieved eTICI 2c or 3
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | SR Classic | SR Combination | Direct Aspiration
Number analyzed (Participants) | 145 | 414 | 313
Minutes | 29.17 (19.3) | 31.26 (17.5) | 27.05 (19.2)

9. Other Pre Specified Outcome: Safety Outcomes
Description: Prespecified safety outcome measures include all-cause mortality and stroke-related mortality up to 90 days (±14), device and/or procedure related SAEs up to 90 Days (±14), neurological deterioration at 24 hours post procedure, embolization to new territory adjudicated by core lab. and neurological deterioration at 24 hours post-procedure to 48 hours
Time Frame: 90 Days (+/- 14 Days)
Population: The analysis population for each variable determined by available imaging data from the Core Lab
Measure: Count of Participants; unit: Participants
Arm/Group | SR Classic | SR Combination | Direct Aspiration
Number analyzed (Participants) | 247 | 697 | 548
Participants
  All-cause Mortality at 90 days (±14 days) | 28 | 105 | 76
  Stroke-related Mortality at 90 days (±14 days) | 19 | 63 | 38
  Device and/or procedure related SAEs at 90 days (±14 days) | 16 | 40 | 23
  Embolization to New Territory during procedure (Core Lab): number analyzed (Participants) | 245 | 692 | 545
  Embolization to New Territory during procedure (Core Lab) | 2 | 6 | 3
  Symptomatic ICH up to 48 hrs post-procedure | 5 | 15 | 14
  Neurological Deterioration (4 or greater increase in NIHSS) up to 48 hrs post-procedure | 13 | 52 | 47
  Access Site Complications up to 48 hrs post-procedure | 3 | 10 | 2

ADVERSE EVENTS:
Time Frame: 90 Days (+/- 14 Days)
Arm/Group | SR Classic | SR Combination | Direct Aspiration
All-Cause Mortality (participants affected / at risk) | 28/247 | 105/697 | 76/548
Serious Adverse Events (participants affected / at risk) | 69/247 | 220/697 | 176/548
Other Adverse Events (participants affected / at risk) | 26/247 | 44/697 | 27/548
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SR Classic (N=247) | SR Combination (N=697) | Direct Aspiration (N=548)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 6 (6) | 6 (6)
Hyperchromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 4 (4) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 3 (3) | 4 (4)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Cardiac arrest (Cardiac disorders) | 2 (2) | 5 (6) | 5 (5)
Cardiac failure (Cardiac disorders) | 1 (1) | 2 (2) | 6 (6)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 2 (2) | 4 (4)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 4 (4) | 0 (0)
Cardiorenal syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Degenerative mitral valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 7 (7) | 12 (12)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 7 (7) | 10 (10)
General physical health deterioration (General disorders) | 0 (0) | 4 (4) | 2 (2)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vascular stent stenosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular stent thrombosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Corona virus infection (Infections and infestations) | 0 (0) | 2 (2) | 5 (5)
Endocarditis (Infections and infestations) | 3 (3) | 2 (2) | 2 (2)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 13 (13) | 7 (7)
Pneumonia escherichia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 5 (5) | 7 (7)
Septic shock (Infections and infestations) | 1 (1) | 5 (5) | 2 (2)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Systemic candida (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3) | 7 (7)
Urosepsis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Brain herniation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Cerebral artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (1)
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 5 (5) | 0 (0)
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
NIH stroke scale score increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Adult failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Aphasia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Basal ganglia infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Brain compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 8 (8) | 22 (22)
Carotid artery aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Carotid artery dissection (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebellar stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral artery embolism (Nervous system disorders) | 8 (8) | 5 (5) | 4 (4)
Cerebral artery occlusion (Nervous system disorders) | 1 (1) | 1 (1) | 2 (3)
Cerebral artery perforation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral circulatory failure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2) | 8 (8) | 6 (6)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 11 (11) | 7 (7)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 15 (15) | 6 (6)
Haemorrhagic transformation stroke (Nervous system disorders) | 3 (3) | 4 (4) | 13 (13)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Hemiplegia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Intracranial artery dissection (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Intracranial mass (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3)
Monoplegia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neurological decompensation (Nervous system disorders) | 1 (1) | 3 (3) | 9 (9)
Neurological symptom (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 2 (2) | 6 (6)
Stroke in evolution (Nervous system disorders) | 10 (10) | 19 (19) | 13 (13)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 6 (6) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vasogenic cerebral oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (3)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal artery occlusion (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatic haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7) | 13 (13)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 9 (9) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 6 (6)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 8 (8) | 12 (12)
Disability (Social circumstances) | 0 (0) | 1 (1) | 0 (0)
Endarterectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Endotracheal intubation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Intestinal resection (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Medical device implantation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Medical device removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Thyroidectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Vena cava filter insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Aortic thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 3 (3) | 5 (5)
Femoral artery aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 2 (2) | 2 (2)
Reperfusion injury (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular dissection (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Vasospasm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vessel perforation (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SR Classic (N=247) | SR Combination (N=697) | Direct Aspiration (N=548)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 2 (2)
Vessel puncture site thrombosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular access site bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular access site complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular access site discharge (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Carotid artery perforation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 2 (2) | 3 (3) | 4 (4)
Cerebral artery perforation (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral vasoconstriction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 6 (6) | 3 (4) | 2 (2)
Haemorrhagic transformation stroke (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Intracranial artery dissection (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Neurological decompensation (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Stroke in evolution (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 5 (5) | 13 (13) | 3 (3)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vascular dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vasospasm (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/91/NCT03845491/Prot_SAP_000.pdf